CLINICAL TRIAL: NCT06510530
Title: Efficacy and Safety of Astragalus for Symptomatic Alleviation in Patients With High-grade Lymphoma Treated With Chemotherapy: a Double-blind Randomized Placebo-controlled Trial
Brief Title: Astragalus for Symptomatic Alleviation in High-grade Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNZ-0036-24
Record Dates: First submitted 2024-06-30; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-06

CONDITIONS: High-grade Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Astragalus (Experimental)
  Interventions: Dietary Supplement: Astragalus
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astragalus — Patients in the intervention group will receive capsules of the Astragalus plant (scientific name: Astragalus membranaceus, common name: Huang Qi) at an initial dose of 2 grams (4 capsules) per day with the option of increasing the dose to 4 grams (8 capsules) per day according to researchers' assessment and patient tolerance. The dose was determined by a focus group of 5 herbalists and according to data from the literature on oncology patients. The duration of the treatment will be up to a month from the end of the chemotherapy treatment which usually lasts up to six months.
  Arms: Astragalus
Dietary Supplement: Placebo — Placebo capsules that look similar to Astragalus capsules will be given to patients from the control group, between 4 and 8 capsules per day according to the researcher's assessment and tolerability. The duration of the treatment will be up to a month from the end of the chemotherapy treatment which usually lasts up to six months.
  Arms: Placebo

SUMMARY:
Lymphoma is a malignant disease of the lymph nodes. There are different types of lymphoma: when some of the lymphomas are indolent and require only follow-up, in cases of aggressive lymphoma or indolent lymphoma with a burden of disease, treatment is necessary, which usually includes chemotherapy with or without biological drugs. These drugs often cause significant damage to the quality of life, various symptoms including exhaustion, neuropathic pain, nausea/vomiting, cognitive decline, as well as a drop in blood counts with serious life-threatening infections that cause a delay in the treatment date that may affect the prognosis.

Drug treatments for symptomatic relief and improvement in quality of life in patients with lymphoma are missing, with only a partial effect and involving side effects.

Astragalus (scientific name: Astragalus membranaceus, common name: Huang Qi) is a perennial flowering plant common in China with a long history of use in traditional Chinese medicine. It is given in various forms of root in combination with other herbs, medicinal soups and as tablets, capsules, solutions, ointments for local use, or subcutaneous or intravenous injection. In patients with oncological diseases, a systematic review (4 trials on a total of 342 patients) showed an improvement in nausea and vomiting as well as in the immune system in patients with colon cancer who received Chemotherapy. A meta-analysis of 27 studies on 1,843 patients with colon cancer also demonstrated a reduction in chemotherapy-induced nausea in patients who received a combination of astragalus with chemotherapy compared to chemotherapy alone. In another meta-analysis that included 45 trials on 3,236 patients with liver cancer, an improvement in 12-month survival was reported with products containing astragalus. In a randomized study of 136 patients with lung cancer, three treatment cycles with astragalus by injection in combination with chemotherapy (vinorelbine and cisplatin) resulted in a significant improvement in quality of life compared to the control group that received chemotherapy alone. Similar results found in 23 patients with metastatic malignancy receiving astragalus by injection in combination with chemotherapy. In addition, a study on 90 patients with advanced cancer showed an improvement in fatigue in patients who received astragalus. Also, a pilot study on 60 patients with breast cancer showed that intravenous administration of astragalus improved blood counts in patients who received it in combination with chemotherapy compared to chemotherapy alone. In patients with hematological malignancies, a study was conducted on 498 patients with acute myeloid leukemia and showed that the use of astragalus or plants containing astragalus was associated with improved survival compared to patients who did not receive it. In the context of lymphoma, a pharmacological study in vivo on animals with lymphoma showed that a combination of an astragalus-containing formula with adriamycin-type chemotherapy improved the effect of adriamycin for the treatment of B-cell lymphoma. Another study in patients who had completed conventional chemotherapy with Rituximab Cyclophosphamide Adriamycine Vincristine Prednisone (R-CHOP) for diffuse large B-cell lymphoma showed that administration of a formula containing astragalus improved immune function and blood counts. Finally, a randomized placebo-controlled study showed that giving a formula containing astragalus to patients under R-CHOP chemo-immunotherapy as first line for diffuse large B cell lymphoma high risk significantly reduced the appearance of side effects from the treatment and improved response to the treatment chemotherapy compared to the control group.

Side effects attributed to astragalus include fatigue, weakness, headaches and hypotension, but in the cited studies and meta-analyses, no increase in the rate of side effects was found in the groups of patients who received this plant compared to the control groups, and no safety problems were described in the use of astragalus in combination with chemotherapy.

In light of the multitude of symptoms that affect the quality of life and adherence to treatment in patients with lymphoma receiving chemotherapy, and in light of the encouraging findings in the literature about symptomatic improvement as a result of combining astragalus during chemotherapy in various malignancies, the investigators aim to examine the effectiveness and safety of astragalus during the treatment of patients with high-grade lymphoma on symptomatic relief and adherence to chemotherapy in a randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Diagnosis of high-grade lymphoma
* Need to start treatment for lymphoma that includes chemotherapy as first line
* Possibility to answer questionnaires once a month
* Signing an informed consent form

Exclusion Criteria:

* Taking up to a week before the randomization a drug with the potential for an interaction of major clinical significance with Astragalus according to a professional database
* Administration of chemotherapy in the past
* Significant disturbance in liver enzymes: Aspartate transaminase and/or alanine transaminase above 5 times the upper limit of normal
* Significant renal dysfunction: glomerular filtration rate under 30 ml/min according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Active autoimmune disease
* Pregnancy or breastfeeding
* Active participation in another interventional study
* Psychiatric disorder with impaired cognitive qualifications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Quality-of-life | From baseline to end-of-treatment, up to 6 months
  European Organization Research for Treatment of cancer core quality of life (EORTC-QLQ-C30) questionnaire summary score which is calculated from the mean of 13 of the 15 quality-of-life (QLQ-C30) scales of the questionnaire = (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ 100-Fatigue+ 100-Pain+ 100-Nausea_Vomiting+ 100-Dyspnoea+ 100-Sleeping Disturbances+ 100-Appetite Loss+ 100-Constipation+ 100-Diarrhoea)/13. Scores range from minimum 0 to maximum 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

SECONDARY OUTCOMES:
Symptoms | From baseline to end-of-treatment, up to 6 months
  Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire at end of treatment: two main concerns of the patient which are rated for severity using a simple numerical Likert scale 0-6 (0: not concerning at all; 6: very concerning).
Fatigue | From baseline to end-of-treatment, up to 6 months
  European Organization Research for Treatment of cancer core quality of life (EORTC-QLQ-C30) questionnaire fatigue score. Scores range from minimum 0 to maximum 100; a higher score represents a higher ("worse") level of fatigue.

OTHER OUTCOMES:
Nausea and vomiting | From baseline to end-of-treatment, up to 6 months
  European Organization Research for Treatment of cancer core quality of life (EORTC-QLQ-C30) questionnaire nausea&vomiting score. Scores range from minimum 0 to maximum 100; a higher score represents a higher ("worse") level of nausea and vomiting.
Cognitive function | From baseline to end-of-treatment, up to 6 months
  European Organization Research for Treatment of cancer core quality of life (EORTC-QLQ-C30) questionnaire cognitive functioning score. Scores range from minimum 0 to maximum 100; a higher score represents a higher ("better") level of cognitive functioning.
Severe neutropenia | Evaluated at day 10-13 of each cycle (each cycle is 14-28 days depending on chemotherapy protocol) during the study treatment (up to 6 months)
  Frequency of severe neutropenia episodes defined as absolute neutrophil count under 0.5x10^9/L
Packed cells transfusion | Through the study treatment, up to 6 months
  Frequency of packed cells transfusion during the study treatment
Use of Granulocyte colony stimulating factors (G-CSF) | Through the study treatment, up to 6 months
  Frequency of G-CSF use during the study treatment
Infections | Through the study treatment, up to 6 months
  Frequency of infections during the study treatment
Hospitalizations | Through the study treatment, up to 6 months
  Frequency of hospitalizations during the study treatment
Compliance to chemotherapy | Through the study treatment, up to 6 months
  Relative dose intensity (RDI) which is the ratio of delivered dose intensity (DDI) of chemotherapy with standard dose intensity (SDI) of chemotherapy = DDI/SDI
Overall response rate (ORR) | Through the study treatment, up to 6 months
  Percentage of patients who have a partial response or complete response to the treatment of lymphoma
Complete response (CR) rate | Through the study treatment, up to 6 months
  Percentage of patients who have a complete response to the treatment of lymphoma
Progression-free survival (PFS) | Up to 2 years after end-of-study treatment: up to 2.5 years
  The length of time during and after the treatment of lymphoma (first line) that patient lives and disease does not progress
Overall survival (OS) | Up to 2 years after end-of-study treatment: up to 2.5 years
  The length of time during and after the treatment of lymphoma (first line) that patient lives
Incidence of Treatment-Emergent Adverse Events | Through the study treatment, up to 6 months
  According to report of adverse events, severe adverse events, drug interactions
Economic analysis | Through the study treatment, up to 6 months
  Calculation of quality-adjusted life years based on EuroQol-5 Dimension (EQ-5D) scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient indicates health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ visual analogue scale (VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Levy Yurkovski, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT06510530/Prot_SAP_000.pdf